CLINICAL TRIAL: NCT04457440
Title: A Pilot Study of a Cognitive Behavioral Sleep Intervention for the Prevention of Type 2 Diabetes
Brief Title: Cognitive Behavioral Sleep Intervention for Prevention of Type 2 Diabetes
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID pandemic affected recruitment.
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Dr. Chan Wai Sze, Assistant Professor, The University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: EA1909037; UW20-245 (Other: HKU/HA HKW IRB)
Record Dates: First submitted 2020-06-26; First posted 2020-07-07 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-10

CONDITIONS: PreDiabetes; Insomnia; Sleep Deprivation
Keywords: Cognitive Behavioral Therapy; Lifestyle Intervention
MeSH Terms: conditions — Prediabetic State; Sleep Initiation and Maintenance Disorders; Sleep Deprivation

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intensive Lifestyle Intervention (ILI) (Active Comparator): The ILI will consist of 8 group-based 90-min sessions focusing on modifying dietary and exercise habits with the goal of reducing 450kcal of daily calories and increasing physical activity to 150 minutes of exercise per week.
  Interventions: Behavioral: Intensive Lifestyle Intervention
- ILI enhanced with cognitive behavioral sleep intervention (Experimental): The ILI+Sleep intervention will consist of the same 8 sessions of ILI with additions of sleep components in each session.
  Interventions: Behavioral: Intensive Lifestyle Intervention enhanced with Cognitive Behavioral Sleep Intervention

INTERVENTIONS:
Behavioral: Intensive Lifestyle Intervention — This intervention is an abbreviated version of the Diabetes Prevention Program, which has been shown to be effective in reducing the risk of developing type 2 diabetes.
  Arms: Intensive Lifestyle Intervention (ILI)
Behavioral: Intensive Lifestyle Intervention enhanced with Cognitive Behavioral Sleep Intervention — This intervention will consist of the same 8 sessions of ILI with additions of sleep components in each session. The additional sleep components will include (a) psychoeducation about the importance of sleep in weight control and glycemic control, (b) sleep hygiene, (c) stimulus control, (d) modifying maladaptive beliefs about sleep, (e) and, setting individualized sleep schedule and reviewing sleep schedule.
  Arms: ILI enhanced with cognitive behavioral sleep intervention

SUMMARY:
The proposed study aims to evaluate if improving sleep could enhance the intensive lifestyle intervention for improving weight loss and glycemic control in prediabetic individuals who have insomnia with short sleep duration. A cognitive behavioral intervention for insomnia with adjustments aimed at increasing sleep duration (CBT-Sleep) will be used for this study.

ELIGIBILITY:
Inclusion Criteria:

* (a) Hong Kong residents,
* (b) BMI > 23kg/m2,
* (c) aged 18 to 65 year-old,
* (d) have prediabetes, defined by a plasma fasting glucose concentration of 5.6 to 6.9 mmol/L, impaired glucose tolerance (2hglucose 7.8-11.0 on OGTT), or HbA1c 5.7-6.4%,
* (e) have average habitual sleep duration < 6.5 hours, confirmed by actigraphy measure of sleep for 2 weeks or have insomnia, confirmed in a clinical sleep interview and actigraph-measure of greater than 30 minutes of sleep onset latency or nighttime awakening for 3 nights or more per week

Exclusion Criteria:

* (a) have unmanaged sleep apnea or other sleep disorders,
* (b) have any current severe mental illnesses,
* (c) have any medical conditions or medication use that could undermine the efficacy of the sleep intervention,
* (d) have shift work schedules,
* (e) have any environmental constraints on the feasibility of implementing a sleep schedule of at least 7.5 hours

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2020-07-01 (Actual); Primary Completion 2021-12-30 (Estimated); Study Completion 2021-12-30 (Estimated)

PRIMARY OUTCOMES:
Changes in HbA1C (%) | 12 weeks from baseline
Changes in fasting glucose concentration (mg/dl) | 12 weeks from baseline
Changes in 2-hr oral glucose tolerance (mg/dl) | 12 weeks from baseline

SECONDARY OUTCOMES:
Changes in insomnia symptom severity | 12 weeks from baseline
  measured by the Insomnia Severity Index. The score ranges from 0 to 28. The higher the score, the greater the symptom severity
Changes in subjective sleep onset latency | 12 weeks from baseline
  measured by daily sleep diary
Changes in subjective wake after sleep onset | 12 weeks from baseline
  measured by daily sleep diary
Changes in subjective total sleep time | 12 weeks from baseline
  measured by daily sleep diary
Changes in objective sleep onset latency | 12 weeks from baseline
  measured by actigraphy
Changes in objective wake after sleep onset | 12 weeks from baseline
  measured by actigraphy
Changes in objective total sleep time | 12 weeks from baseline
  measured by actigraphy
Changes in body weight (kg) | 12 weeks from baseline
Changes in psychological distress | 12 weeks from baseline
  the validated Chinese version of the Depression Anxiety Stress Scales (DASS-21)will be used. The score ranges from 0 to 63. The higher the score, the greater the distress
Changes in quality of life | 12 weeks from baseline
  the validated Chinese version of the Satisfaction with Life Scale will be used to measure quality of life. The score ranges from 5 to 35. The higher the score, the greater the quality of life
Changes in food craving | 12 weeks from baseline
  Measured by the Food Craving Questionnaire. The score ranges from 10 to 70. The higher the score, the greater the food craving
Changes in acceptance of physical activity | 12 weeks from baseline
  Measured by the Physical Activity Acceptance and Action Questionnaire. The score ranges from 10 to 70. The higher the score, the greater acceptance.
Changes in weight loss self efficacy | 12 weeks from baseline
  Measured by the Weight Loss Self Efficacy Scale. The score ranges from 0 to 100%. The higher the percentage, the greater the self-efficacy
Changes in weight control strategies | 12 weeks from baseline
  Measured by the Weight Control Strategy Scale. The score ranges from 0 to 120. The higher the percentage, the more effective strategies are used
Changes in dietary composition | 12 weeks from baseline
  Measured by the Chinese version of the 7-day Food Frequency Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Wai Sze Chan, PhD, Principal Investigator — The University of Hong Kong
Locations (2):
- Hong Kong (2):
  - Queen Mary Hpspital, Hong Kong
  - The University of Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Deidentified data will be shared with other researchers for review purposes.
Supporting Information: Study Protocol, SAP